CLINICAL TRIAL: NCT05240703
Title: Efficacy of Stabilization Splint Treatment on Facial Pain - One-year Follow-up
Brief Title: Stabilization Splint Treatment of TMD
Acronym: TMD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oulu (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 29/2007
Record Dates: First submitted 2022-01-20; First posted 2022-02-15 (Actual); Last update posted 2022-02-15 (Actual); Status verified 2022-02

CONDITIONS: Temporomandibular Disorder; Facial Pain
Keywords: temporomandibular disorders; TMD; facial pain; treatment; stabilization splint; clinical trial
MeSH Terms: conditions — Temporomandibular Joint Disorders; Facial Pain

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: The same dentist examiner conducted all of the follow-up examinations, being unaware of the group status of the patients.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stabilization splint group (Experimental): The patients in the splint group were treated with a stabilization splint and received counseling and instructions for masticatory muscle exercises
  Interventions: Device: Stabilization splint treatment
- Control group (No Intervention): The controls received only counseling and instructions for masticatory muscles exercises.

INTERVENTIONS:
Device: Stabilization splint treatment — The stabilization splints were made of heat-cured acrylic by the same dental technician. The occlusion of the splint was defined in the centric relation occlusion using wax (Astynax, Associated Dental Products Ltd, UK). The patients were instructed to use the splint every night during the course of the study. The patients were instructed to perform a standardized program for masticatory muscle exercises. At the beginning of the training program, active mouth openings, laterotrusive movements and protrusive movements were performed. The mandible was held in the maximal positions for a few seconds on each movement. Thereafter, these movements were made towards resistance (using the patient's own fingers). After jaw exercises, the patients were suggested to open the jaw wide, stretching it with fingers a few times for 10 to 20 seconds. These movements were repeated 7 to 10 times per training session, and the sessions were performed 2-3 times per day.
  Arms: Stabilization splint group

SUMMARY:
The aim of this randomized controlled trial was to assess the efficacy of stabilization splint treatment on TMD-related facial pain and oral health-related quality of life during a one-year follow-up. Eighty TMD patients were randomly assigned to two groups: splint group (n=39) and control group (n=41). The patients in the splint group were treated with a stabilization splint and received counseling and instructions for masticatory muscle exercises. The controls received only counseling and instructions for masticatory muscles exercises.

The outcome variables were the intensity of facial pain (as measured with visual analogue scale, VAS), patients' subjective estimate of symptoms and treatment outcome, as well as Oral Heath Impact Profile (OHIP)-14. The differences in variables between the groups at each follow-up points (1 month, 3 months, 6 months and 1 year after baseline) were analyzed using regression models. Group status and presence of psychosocial symptoms were included as the explanatory factor and baseline VAS, gender, age, length of treatment and general health status as confounders.

DETAILED DESCRIPTION:
DESIGN OF THE STUDY The study sample consisted originally of 80 patients (18 men, 62 women) who were referred to the Oral and Maxillofacial Department in Oulu University Hospital, Oulu, Finland, for treatment of TMD-related facial pain. The patients were examined between March 2008 and August 2010. The inclusion criteria were the following: 1. clinically diagnosed TMD as defined by the Research Diagnostic Criteria for Temporomandibular Disorders (RDC/TMD) (1), 2. minimum of 20 years of age and 3. lack of long-term illnesses (i.e. rheumatoid arthritis) that may affect TMJs or the masticatory muscles.

Using computer generated random numbers, the patients were randomly assigned to two groups: splint group and control group. Patients in the control group (n=41) were given counseling and guidance for masticatory muscle exercises. In addition to these, the patients in the splint group (n=39) were also treated with a stabilization splint.

DATA COLLECTION The patients had four follow-ups: at about 1 month, 3 months, 6 months and one year after the baseline evaluation. The same dentist specialized in stomatognathic physiology (KS) conducted all of the follow-up examinations, being unaware of the group status of the patients. At baseline the psychosocial screening (depression symptoms, non-specific physical symptoms, pain-related disability) was performed using RDC/TMD Axis II instruments. At baseline and at all the follow-ups the intensity of the facial pain was assessed using Visual Analogue Scale (VAS). The patients' subjective estimates of the effects of the treatment were evaluated with a questionnaire, using a scale from 1 to 4 (1= Very good effect, 2= Treatment has helped to some extent, 3= No difference / Cannot tell and 4= Symptoms worsened). The patients' general health status was also inquired by a questionnaire (on a scale of 1-5, 1=excellent, 2=very good, 3=good, 4=moderate, 5=poor). The patients filled in the Oral Health Impact Profile-14 (OHIP-14) questionnaire before treatment and at 3 months, 6 months and 1 year.

TREATMENT PROCEDURES The stabilization splints were made of heat-cured acrylic by the same dental technician. The occlusion of the splint was defined in the centric relation occlusion using wax (Astynax, Associated Dental Products Ltd, UK). The patients were instructed to use the splint every night during the course of the study.

All the patients in both groups were instructed to perform a standardized program for masticatory muscle exercises as described by Carlsson and Magnusson (1992). At the beginning of the training program, active mouth openings, laterotrusion and protrusion movements were performed. The mandible was held in the maximal positions for a few seconds on each movement. Thereafter, these movements were made towards resistance (using the patient's own fingers). After jaw exercises, the patients were suggested to open the jaw wide, stretching it with fingers a few times for 10 to 20 seconds. These movements were repeated 7 to 10 times per training session, and the sessions were performed 2-3 times per day. The patients received written instructions, and the movements were also demonstrated by the dentist before the treatment, and reprised if necessary. The instructions for masticatory muscle exercises were given by the same dentist (KS) at the first visit. At every examination the patients were reminded to use the splint and/or to perform the exercises at a regular basis.

The stabilization splint treatments were performed by two other dentists who were instructed in the treatment method.

ATTRITION All of the patients in the total sample were defined as belonging to the "intention-to-treat" (ITT) population. Thus, the ITT also included those who switched groups or those who in whichever group received other treatment than initially planned based on the group criteria. In the analysis, the number of days each patient had stayed in the assigned groups was taken into account. The patients who had stayed in their assigned groups for the whole follow-up period were defined as forming the "per-protocol" (PP) population.

STATISTICAL ANALYSIS Statistical significances of the differences in patients' estimate of the effects of the treatment between the groups were analyzed using chi-square test. Differences in means of the change in VAS between the groups were tested using ANOVA. VAS change was calculated by subtracting VAS at one-year follow-up from baseline VAS. The fluctuation of facial pain during the study (VAS) was demonstrated with a box-plot diagram. At first, linear regression analysis was used to analyze factors associated with change in VAS after one-year follow-up in both the ITT and PP populations. Group status was included as the explanatory factor and baseline VAS, gender, age, length of treatment and general health status were included as confounders. Linear mixed-effect regression model was used to analyse factors associated with change in OHIP severity during the 1-year follow-up, taking into account treatment time, age, gender and group status. The effect of depression and non-specific physical symptoms on the intensity of facial pain, as measured with visual analogue scale (VAS) was estimated with linear mixed models.

ELIGIBILITY:
Inclusion Criteria

* clinically diagnosed TMD according to the RDC/TMD
* age > 20 years

Exclusion Criteria:

• Presence of any chronic diseases, such as rheumatoid arthritis, that may affect the TMJ or the masticatory muscles

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2008-03-01 (Actual); Primary Completion 2010-08-31 (Actual); Study Completion 2010-08-31 (Actual)

PRIMARY OUTCOMES:
Change in facial pain intensity | from baseline to 1-year follow-up
  The change of the intensity of the facial pain, assessed using Visual Analogue Scale (VAS) on a 0 (no pain) to 10 (pain as bad as could be) rating
Subjective estimate on treatment outcome | 1 month follow-up
  The patients' subjective estimates of the effects of the treatment were evaluated with a questionnaire, using a scale from 1 to 4 (1= Very good effect, 2= Treatment has helped to some extent, 3= No difference / Cannot tell and 4= Symptoms worsened).
Subjective estimate on treatment outcome | 3 month follow-up
  The patients' subjective estimates of the effects of the treatment were evaluated with a questionnaire, using a scale from 1 to 4 (1= Very good effect, 2= Treatment has helped to some extent, 3= No difference / Cannot tell and 4= Symptoms worsened).
Subjective estimate on treatment outcome | 6 month follow-up
  The patients' subjective estimates of the effects of the treatment were evaluated with a questionnaire, using a scale from 1 to 4 (1= Very good effect, 2= Treatment has helped to some extent, 3= No difference / Cannot tell and 4= Symptoms worsened).
Subjective estimate on treatment outcome | 1 year follow-up
  The patients' subjective estimates of the effects of the treatment were evaluated with a questionnaire, using a scale from 1 to 4 (1= Very good effect, 2= Treatment has helped to some extent, 3= No difference / Cannot tell and 4= Symptoms worsened).
Subjective estimate on symptom severity | 1 month follow-up
  The subjective assessment of the severity of TMD symptoms after treatment was assessed by means of a scale on 1 to 5 (1= 'no symptoms'/ 'symptoms not significant', 2 = 'mild symptoms', 3 = 'moderate symptoms', 4 = 'severe symptoms', 5 = 'intolerable symptoms')
Subjective estimate on symptom severity | 3 month follow-up
  The subjective assessment of the severity of TMD symptoms after treatment was assessed by means of a scale on 1 to 5 (1= 'no symptoms'/ 'symptoms not significant', 2 = 'mild symptoms', 3 = 'moderate symptoms', 4 = 'severe symptoms', 5 = 'intolerable symptoms')
Subjective estimate on symptom severity | 6 month follow-up
  The subjective assessment of the severity of TMD symptoms after treatment was assessed by means of a scale on 1 to 5 (1= 'no symptoms'/ 'symptoms not significant', 2 = 'mild symptoms', 3 = 'moderate symptoms', 4 = 'severe symptoms', 5 = 'intolerable symptoms')
Subjective estimate on symptom severity | 1 year follow-up
  The subjective assessment of the severity of TMD symptoms after treatment was assessed by means of a scale on 1 to 5 (1= 'no symptoms'/ 'symptoms not significant', 2 = 'mild symptoms', 3 = 'moderate symptoms', 4 = 'severe symptoms', 5 = 'intolerable symptoms')
Change of Oral health related quality of life (OHRQoL) | from baseline to 1-year follow-up
  Change of Oral health related quality of life was assessed using Oral Health Impact Profile (OHIP-14, sum score from 0 to 56, the higher value indicating poorer OHRQoL)

CONTACTS AND LOCATIONS:
Overall Officials: Kirsi Sipilä, Professor, Principal Investigator — Research Unit of Oral Health Sciences, University of Oulu, Finland

REFERENCES:
- [Background] Dworkin SF, LeResche L. Research diagnostic criteria for temporomandibular disorders: review, criteria, examinations and specifications, critique. J Craniomandib Disord. 1992 Fall;6(4):301-55. No abstract available. PMID 1298767
- [Result] Huttunen J, Qvintus V, Suominen AL, Sipila K. Role of psychosocial factors on treatment outcome of temporomandibular disorders. Acta Odontol Scand. 2019 Mar;77(2):119-125. doi: 10.1080/00016357.2018.1511057. Epub 2018 Sep 28. PMID 30264631
- [Result] Kokkola O, Suominen AL, Qvintus V, Myllykangas R, Lahti S, Tolvanen M, Sipila K. Efficacy of stabilisation splint treatment on the oral health-related quality of life-A randomised controlled one-year follow-up trial. J Oral Rehabil. 2018 May;45(5):355-362. doi: 10.1111/joor.12622. PMID 29512838
- [Result] Qvintus V, Suominen AL, Huttunen J, Raustia A, Ylostalo P, Sipila K. Efficacy of stabilisation splint treatment on facial pain - 1-year follow-up. J Oral Rehabil. 2015 Jun;42(6):439-46. doi: 10.1111/joor.12275. Epub 2015 Jan 17. PMID 25644634